CLINICAL TRIAL: NCT01926977
Title: Evaluation of Post Injection Inflammation and Pain After Ranibizumab vs Aflibercept Intravitreal Injections
Brief Title: Evaluation of Pain and Inflammation After Injection of Lucentis vs Eylea for Treatment of Wet Macular Degeneration
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Arshad Khanani (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Arshad Khanani, Vitreo-Retinal Surgeon, Sierra Eye Associates
Organization: Sierra Eye Associates (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ML28895; 20131227 (Other: Western Institutional Review Board)
Record Dates: First submitted 2013-08-19; First posted 2013-08-21 (Estimated); Results first posted 2016-03-03 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-02

CONDITIONS: Neovascular Age-Related Macular Degeneration
MeSH Terms: interventions — Ranibizumab; aflibercept

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ranibizumab 0.5mg Intravitreal injection (Active Comparator): Intravitreal injection of Ranibizumab 0.5mg once
  Interventions: Drug: Ranibizumab 0.5mg
- Aflibercept 2.0mg Intravitreal injection (Active Comparator): Intravitreal Aflibercept 2.0mg once
  Interventions: Drug: Aflibercept 2.0mg

INTERVENTIONS:
Drug: Ranibizumab 0.5mg — Patient will receive intravitreal injection of Ranibizumab 0.5mg.
  Other Names: Lucentis
  Arms: Ranibizumab 0.5mg Intravitreal injection
Drug: Aflibercept 2.0mg — Patients will receive intravitreal injection of Aflibercept 2.0mg.
  Other Names: Eylea
  Arms: Aflibercept 2.0mg Intravitreal injection

SUMMARY:
This study is designed to compare the post injection inflammation and pain seen after intravitreal injections of Ranibizumab vs Aflibercept.

DETAILED DESCRIPTION:
This is an open-label, Phase I-II study of post injection pain and inflammation after intravitreally administered Ranibizumab and Aflibercept in 100 subjects with Neovascular Age-Related Macular Degeneration. We will enroll both treatment experienced ( patients who were treated with Lucentis or Eylea, but not Avastin in the past) and treatment naive patients ( new onset Neovascular AMD with no history of intravitreal injections).

The treatment experienced patients will be treated with the intravitreal medication other than what they were receiving in the past, for example, patients treated with Lucentis will switch to Eylea for study purposes and vice versa.

Consented, enrolled subjects will receive open-label intravitreal injection of either 0.5mg Ranibizumab or 2mg Aflibercept. A standard intravitreal injection protocol will be followed. Patients will be reevaluated between 24-48 hours and 5-7 days post injections. A non-injecting physician will evaluate the patients for anterior chamber inflammation; this physician will be blinded about the specific treatment. Anterior chamber inflammation is described as any cell or flare in the anterior chamber. These will be evaluated using Standardization of Uveitis Nomenclature (SUN) working group classifications.

Pain score will be evaluated using a Numerical Rating Scale. Each patient will have a standard script verbally read to them at their visit, and asked to rate their pain based on this scale.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide informed consent and comply with study assessments for the full duration of the study
2. Age >/= 65 years
3. New onset Neovascular Age-Related Macular Degeneration or (See No.4)
4. Previously treated Neovascular Age-Related Macular Degeneration with Lucentis or Eylea intravitreal injections
5. Visual Acuity of 20/400 or better
6. No history of Post injection pain or inflammation with prior treatments -

Exclusion Criteria:

1. History of Endophthalmitis in either eye
2. Uncontrolled or symptomatic Dry Eye Syndrome
3. History of Anterior or Posterior Uveitis
4. History of Post injection pain or inflammation with prior treatments
5. Recent thromboembolic event(<3 months)
6. Pregnancy(positive pregnancy test) or Lactation/Premenopausal women not using adequate contraception -

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-09; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arshad M Khanani, MD, Principal Investigator — Sierra Eye Associates
Locations (1):
- Sierra Eye Associates, Reno, Nevada, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ranibizumab 0.5mg Intravitreal Injection | Aflibercept 2.0mg Intravitreal Injection
Started | 47 | 53
Completed | 47 | 53
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ranibizumab 0.5mg Intravitreal Injection | Aflibercept 2.0mg Intravitreal Injection | Total
Number analyzed (Participants) | 47 | 53 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 47 | 53 | 100
Age, Continuous [Mean (Full Range); unit: years] | 76.3 [65 to 96] | 80.6 [67 to 95] | 78.6 [65 to 96]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 34 | 60
  Male | 21 | 19 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 4 | 4
  Not Hispanic or Latino | 47 | 48 | 95
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 0 | 0 | 0
  White | 46 | 52 | 98
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 47 | 53 | 100

OUTCOME MEASURES:

1. Primary Outcome: Evidence of Anterior Chamber Inflammation
Description: Evidence of anterior chamber inflammation at visit #1 and #2 using Standardization of Uveitis Nomenclature (SUN)
Time Frame: 24 to 48 hours (visit #1) and 5 to 7 days (visit #2)
Measure: Number; unit: participants
Arm/Group | Ranibizumab 0.5mg Intravitreal Injection | Aflibercept 2.0mg Intravitreal Injection
Number analyzed (Participants) | 47 | 53
participants
  Inflammation at visit 1 | 1 | 10
  Inflammation at visit 2 | 0 | 1

2. Secondary Outcome: Patients With Post Injection Pain Score of One or Higher on Pain Scale
Description: Pain score rated on an 11 point numerical rating from 0-10 ( 0 = no pain, and 10 = worst possible pain) administered to each patient verbally at visit #1 and visit #2. The data below shows number of patients with pain score 1 or greater in each group.
Time Frame: 24 to 48 hours (visit #1) and 5 to 7 days (visit #2)
Measure: Number; unit: participants
Arm/Group | Ranibizumab 0.5mg Intravitreal Injection | Aflibercept 2.0mg Intravitreal Injection
Number analyzed (Participants) | 47 | 53
participants
  Subjects with pain score 1 or higher at visit 1 | 7 | 9
  Subjects with pain score 1 or higher at visit 2 | 0 | 1

ADVERSE EVENTS:
Arm/Group | Ranibizumab 0.5mg Intravitreal Injection | Aflibercept 2.0mg Intravitreal Injection
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/53
Other Adverse Events (participants affected / at risk) | 1/47 | 10/53
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ranibizumab 0.5mg Intravitreal Injection (N=47) | Aflibercept 2.0mg Intravitreal Injection (N=53)
Anterior chamber inflammation at Visit 1 (Eye disorders) | 1 (1) | 10 (10) — All patients in this group had 0.5+ inflammation as reported using Standardization of Uveitis Nomenculature working group classification.
Anterior chamber inflammation at Visit 2 (Eye disorders) | 0 (0) | 1 (1) — Patient had 1+ inflammation as reported using Standardization of Uveitis Nomenculature working group classification.
Vitreous inflammation at Visit 1 (Eye disorders) | 0 (0) | 4 (4) — Inflammation was mild and was graded as 0.5 on Nussenblatt scale
Vitreous inflammation at Visit 2 (Eye disorders) | 0 (0) | 1 (1) — Inflammation was mild and was graded as 0.5 on Nussenblatt scale

LIMITATIONS AND CAVEATS:
Small sample size. Non-randomized choice of medications.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes